CLINICAL TRIAL: NCT06743061
Title: Evaluation of Arthroscopic Debridement, Subacromial Decompression, and Biceps Tenotomy Without Repair of Rotator Cuff in Chronic Massive Rotator Cuff Tear
Brief Title: Long-Term Follow-up of Arthroscopic Biceps Tenotomy and Subacromial Decompression in Chronic Massive Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Ghanem, Orthopedic Surgeon, MSc Candidate, Cairo University
Other Study IDs: RC-1911-2018
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group I
  Interventions: Behavioral: Post-Op Follow Up

INTERVENTIONS:
Behavioral: Post-Op Follow Up — Post Arthroscopic Biceps Tenotomy and Subacromial Decompression in Chronic Massive Rotator Cuff Tears.

SUMMARY:
Chronic massive rotator cuff tears (MMRCTs) are a significant orthopedic challenge, often leading to significant shoulder pain and functional impairment. While surgical intervention is a common treatment approach, long-term outcomes and the optimal surgical technique remain debatable. Arthroscopic debridement, subacromial decompression, and biceps tenotomy are frequently employed procedures, but their long-term effectiveness in managing MMRCTs is not fully understood. A comprehensive understanding of the long-term outcomes of these procedures is crucial for guiding clinical decision-making and patient counseling.

The study aims to evaluate the long-term clinical and functional outcomes of arthroscopic debridement, subacromial decompression, and biceps tenotomy in patients with chronic massive rotator cuff tears. By analyzing a cohort of patients who underwent these procedures, we will assess factors influencing long-term outcomes, such as patient demographics, preoperative functional status, and surgical technique. Furthermore, we will compare the long-term results of this surgical approach to other treatment modalities, including open repair and conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had arthroscopic debridement with subacromial decompression and biceps tenotomy without rotator cuff repair for chronic massive Rotator Cuff Tears

Exclusion Criteria:

* Patient who hadn't met the requirements for arthroscopic debridement with subacromial decompression and biceps tenotomy without rotator cuff repair for chronic massive Rotator Cuff Tears

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From Oct 2018 to Jan 2021, 23 patients who had chronic massive RCTs received arthroscopic management for their RCTs and were followed as short-term follow-up for 3 months after surgery. Then, patients were asked to attend the Orthopedic outpatient clinic every three months for assessment to get the outcomes of the long-term follow-up. The preoperative, operative, immediate postoperative, and short-term follow-up data were collected from patients' files.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
The proportion of patients reported having at least a 50% obtaining the normal angle of forward flexion and painless range of movement with approved normal acromiohumeral distance. | 42 Months
  The Success rate of Arthroscopic debridement with subacromial decompression and biceps tenotomy without rotator cuff repair for chronic massive Rotator cuff tear in making the patients able to obtain the normal angle of forward flexion and painless range of movement with approved normal acromiohumeral distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Kasr Al-Einy, Cairo, Egypt